CLINICAL TRIAL: NCT01959347
Title: Effects of Surgical Treatment Enhanced With Exercise for Mixed Urinary Incontinence (ESTEEM)
Brief Title: Combined Treatment for Mixed Incontinence
Acronym: ESTEEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Women and Infants Hospital of Rhode Island (Other); The Cleveland Clinic (Other); Duke University (Other); University of Alabama at Birmingham (Other); University of New Mexico (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); University of California, San Diego (Other); Kaiser Permanente (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFDN-26P01; U10HD041261 (NIH); U10HD069013 (NIH); U10HD054215 (NIH); U10HD041267 (NIH); U10HD054214 (NIH); U10HD069025 (NIH); U10HD069010 (NIH); U10HD041263 (NIH); U01HD069031 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Urinary Incontinence, Stress; Urinary Incontinence, Urge
Keywords: urinary incontinence; midurethral sling; pelvic floor therapy
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Miduretheral Sling (Control) (Sham Comparator): Miduretheral Sling (Control)
  Interventions: Procedure: Miduretheral Sling
- MUS+BPTx (Experimental): Miduretheral Sling with behavioral/pelvic floor therapy
  Interventions: Other: Miduretheral Sling with behavioral/pelvic floor therapy

INTERVENTIONS:
Procedure: Miduretheral Sling — MUS can include the TVT™ (mechanical cut mesh only, Gynecare, ETHICON Women's Health & Urology, Somerville, NJ), TVT-O™ (mechanical cut mesh only, Gynecare), or Monarc™ (American Medical Systems, Minnetonka, MN).
  Other Names: MUS
  Arms: Miduretheral Sling (Control)
Other: Miduretheral Sling with behavioral/pelvic floor therapy — MUS is combined with components of behavioral therapy (designed to change behaviors to encourage continence), and pelvic floor muscle therapy (designed to strengthen the pelvic floor muscles, enhance the physiological closure of the bladder neck, and improve coordination). This is done prior to MUS (1 visit) and after MUS for 5 visits at 2, 4, 6, 8 weeks and 6 months.
  Other Names: MUS + BPTx
  Arms: MUS+BPTx

SUMMARY:
The overarching goal of this randomized trial is to estimate the effect of combined midurethral sling (MUS) and peri-operative behavioral/pelvic floor therapy (BPTx) compared to MUS alone on successful treatment of MUI symptoms in 472 women. Secondary objectives include estimating the effect of combined treatment compared to MUS on improving overactive bladder (OAB) and stress urinary incontinence (SUI) outcomes separately, need for additional treatment, time to failure and identifying predictors of poor outcomes in this MUI population.

A supplemental study, The Human Microbiome Study of ESTEEM, will evaluate the urinary and vaginal microbiome as it relates to women with MUI, their treatment and unaffected controls.

DETAILED DESCRIPTION:
ESTEEM is a multi-center randomized trial of 472 women with MUI who have elected to undergo surgical treatment for SUI. Participants will be randomized to a peri-operative BPTx program+MUS versus MUS alone. The purpose is to compare combined MUS+BPTx versus MUS alone (control) on improving MUI symptoms at 1 year.

Patients will be assigned to one of the two treatment groups. Randomization will be stratified by clinical site and by UUI "severity," which will be defined by the number of urgency urinary IEs on diary.

The primary outcome for this study is the mean change from baseline in UDI-total score at 1 year postoperative. The UDI is a validated, disease-specific, patient-reported outcome (PRO) measure.

Secondary outcomes UUI/OAB outcomes will be measured using the UDI-irritative subscale that measures symptom burden, impact, and changes related to OAB. It is highly responsive to treatment-related change and is able to discriminate among levels of change in all bladder diary variables (urinary urgency, frequency and urge incontinence) and patient ratings of treatment benefit that will characterize how MUS may affect all OAB symptoms individually and as a whole. SUI symptom outcomes will be measured using the UDI-stress subscale to compare SUI outcomes between women randomized to MUS + BPTx versus MUS alone.

Other UUI/OAB outcomes that will be compared between groups include 1) the change in IE frequency and type, number of urgency episodes, urgency severity with voids, number of diurnal voids, and number of nocturnal voids using a bladder diary; 2) patient satisfaction with treatment using the OAB-SAT-q; 3) bother and heal related quality of life using the OAB-q subscale

For analyzing time to failure, "failure" will be defined as initiation of any additional treatment for either SUI or UUI/OAB symptoms during the follow-up period. Subjects lost to follow up will be censored at the time of their last visit.

Quality of life/global impression will be assessed be compared between treatment groups using the a) Incontinence Impact Questionnaire (IIQ), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ), c) European Quality of Life-5 Dimensions (EQ-5D), d) Adaptation Index and e) Patient Global Impression of Improvement (PGI-I) and Patient Global Impression of Severity (PGI-S).

Safety/additional treatments will be characterized as a) additional re-treatments for SUI or UUI within 12 months of treatment, and type of re-treatment and b) return to OR for sling revision due to worsened OAB symptoms.

To evaluate the association between PFM strength and improvements in UI symptoms, we will objectively assess PFM strength changes using the Peritron Perineometer, and instrument specifically designed for pelvic floor assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of both SUI and UUI on bladder diary; and > 2 IEs/3 days

   1. > 1 Stress IE/3 day diary
   2. > 1 Urge IE/3 day diary
2. Reporting at least "moderate bother" from UUI item on the UDI "Do you usually experience urine leakage associated with a feeling of urgency, that is a strong sensation of needing to go to the bathroom?"
3. Reporting at least "moderate bother" from SUI item on UDI "Do you usually experience urine leakage related to coughing, sneezing, or laughing"
4. Diagnosis of SUI defined by a positive cough stress test (CST) or urodynamic evaluation within the past 18 months
5. Desires surgical treatment for SUI symptoms
6. Urinary symptoms >3 months
7. Subjects understand that BPTx is a treatment option for MUI outside of ESTEEM study protocol
8. Urodynamics within past 18 months

Exclusion Criteria:

1. Anterior or apical compartment prolapse at or beyond the hymen (>0 on POPQ), regardless if patient is symptomatic

   a)Women with anterior or apical prolapse above the hymen (<0) who do not report vaginal bulge symptoms will be eligible
2. Planned concomitant surgery for anterior vaginal wall or apical prolapse > 0

   a)Women undergoing only rectocele repair are eligible
3. Women undergoing hysterectomy for any indication will be excluded
4. Active pelvic organ malignancy
5. Age <21 years
6. Pregnant or plans for future pregnancy in next 12 months, or within 12 months post-partum
7. Post-void residual >150 cc on 2 occasions, or current catheter use
8. Participation in other trial that may influence results of this study
9. Unevaluated hematuria
10. Prior sling, synthetic mesh for prolapse, implanted nerve stimulator for incontinence
11. Spinal cord injury or advanced/severe neurologic conditions including Multiple Sclerosis, Parkinsons
12. Women on anti-muscarinic therapy will be eligible after 3 week wash-out period
13. Non-ambulatory
14. History of serious adverse reaction to synthetic mesh
15. Not able to complete study assessments per clinician judgment, or not available for 12 month follow-up
16. Women who only report "other IE" on bladder diary, and do not report at minimum 1 stress and 1 urge IE/3 days
17. Diagnosis of and/or history of bladder pain or chronic pelvic pain
18. Women who had intravesical Botox injection within the past 12 months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-10-28; Primary Completion 2017-08-09 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian W. Sung, Principal Investigator — Brown/ Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery; Dennis Wallace, Principal Investigator — RTI International
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Department of Obstetrics and Gynecology, Birmingham, Alabama
  - Kaiser Permanente -- Downey, Downey, California
  - University of California at San Diego, UCSD Women's Pelvic Medicine Center, La Jolla, California
  - Kaiser Permanente -- San Diego, San Diego, California
  - University of New Mexico Health Sciences Center, Department of Obstetrics and Gynecology, Albuquerque, New Mexico
  - Duke University, Duke Division of Urogynecology and Reconstructive Pelvic Surgery, Durham, North Carolina
  - Cleveland Clinic, Department OB/GYN, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Department of Obstetrics and Gynecology, Pittsburgh, Pennsylvania
  - Brown/ Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richter HE, Carnes MU, Komesu YM, Lukacz ES, Arya L, Bradley M, Rogers RG, Sung VW, Siddiqui NY, Carper B, Mazloomdoost D, Dinwiddie D, Gantz MG; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Association between the urogenital microbiome and surgical treatment response in women undergoing midurethral sling operation for mixed urinary incontinence. Am J Obstet Gynecol. 2022 Jan;226(1):93.e1-93.e15. doi: 10.1016/j.ajog.2021.07.008. Epub 2021 Jul 21. PMID 34297969
- [Derived] Sung VW, Richter HE, Moalli P, Weidner AC, Nguyen JN, Smith AL, Dunivan G, Ridgeway B, Borello-France D, Newman DK, Mazloomdoost D, Carper B, Gantz MG; NICHD Pelvic Floor Disorders Network. Characteristics Associated With Treatment Failure 1 Year After Midurethral Sling in Women With Mixed Urinary Incontinence. Obstet Gynecol. 2021 Aug 1;138(2):199-207. doi: 10.1097/AOG.0000000000004444. PMID 34237755
- [Derived] Sung VW, Richter HE, Moalli P, Weidner AC, Nguyen JN, Smith AL, Dunivan G, Ridgeway B, Borello-France D, Newman DK, Mazloomdoost D, Carper B, Gantz MG; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network*. Characteristics Associated With Treatment Failure 1 Year After Midurethral Sling in Women With Mixed Urinary Incontinence. Obstet Gynecol. 2020 Sep;136(3):482-491. doi: 10.1097/AOG.0000000000003989. PMID 32769647 (Retraction: PMID 34293762 Obstet Gynecol. 2021 Aug 1;138(2):312)
- [Derived] Sung VW, Borello-France D, Newman DK, Richter HE, Lukacz ES, Moalli P, Weidner AC, Smith AL, Dunivan G, Ridgeway B, Nguyen JN, Mazloomdoost D, Carper B, Gantz MG; NICHD Pelvic Floor Disorders Network. Effect of Behavioral and Pelvic Floor Muscle Therapy Combined With Surgery vs Surgery Alone on Incontinence Symptoms Among Women With Mixed Urinary Incontinence: The ESTEEM Randomized Clinical Trial. JAMA. 2019 Sep 17;322(11):1066-1076. doi: 10.1001/jama.2019.12467. PMID 31529007

RESULTS

PARTICIPANT FLOW:
Groups:
- MUS Only: Midurethral sling alone
- MUS+BPTx: Midurethral sling and behavioral/pelvic floor therapy
Period: Overall Study
Arm/Group | MUS Only | MUS+BPTx
Started | 238 | 242
Completed | 229 | 235
Not Completed | 9 | 7
Not completed — Protocol Violation | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MUS Only | MUS+BPTx | Total
Number analyzed (Participants) | 229 | 235 | 464
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (10.4) | 54.3 (11) | 54 (10.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 229 | 235 | 464
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 3 | 7 | 10
  Asian | 1 | 2 | 3
  Black/African American | 19 | 22 | 41
  More than one race | 1 | 2 | 3
  Other | 23 | 19 | 42
  Unknown/Not Reported | 1 | 2 | 3
  White | 181 | 181 | 362
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latina | 56 | 49 | 105
  Not Hispanic/Not Latina | 169 | 184 | 353
  Unknown/Not Reported | 4 | 2 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (7) | 31.7 (7) | 32 (7)
Current Smoker [Count of Participants; unit: Participants]
  No | 200 | 203 | 403
  Yes | 28 | 32 | 60
  Unknown or Not Reported | 1 | 0 | 1
Ever Pregnant [Count of Participants; unit: Participants]
  No | 10 | 15 | 25
  Yes | 218 | 220 | 438
  Unknown or Not Reported | 1 | 0 | 1
Number of Vaginal Deliveries [Median (Full Range); unit: Number of deliveries] | 2 [0 to 13] | 2 [0 to 7] | 2 [0 to 13]
Number of Cesarean Deliveries [Median (Full Range); unit: Number of deliveries] | 0 [0 to 5] | 0 [0 to 5] | 0 [0 to 5]
Menstrual Status [Count of Participants; unit: Participants]
  not sure | 28 | 32 | 60
  post-menopausal | 124 | 138 | 262
  pre-menopausal | 76 | 65 | 141
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline UDI Total Score
Description: The Urogenital Distress Inventory (UDI) is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI scale has a range from 0 to 300 with higher scores indicating greater distress. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed. Data that was collected after a participant was retreated for urinary incontinence was excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 195
  3 Months | -138.8 [-145.9 to -131.7] | -142.7 [-150.7 to -134.8]
  6 Months: number analyzed (Participants) | 176 | 183
  6 Months | -137 [-145 to -128.9] | -147.4 [-155.4 to -139.4]
  12 Months: number analyzed (Participants) | 174 | 182
  12 Months | -137.9 [-145.9 to -129.8] | -147.7 [-156.4 to -139]

2. Secondary Outcome: Change From Baseline UDI Stress Score
Description: The Urogenital Distress Inventory is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI Stress subscale has a range from 0 to 100 with higher scores indicating greater distress. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 195
  3 Months | -70.6 [-74.1 to -67.1] | -72.5 [-76.4 to -68.6]
  6 Months: number analyzed (Participants) | 176 | 183
  6 Months | -69.5 [-73.8 to -65.2] | -72.8 [-76.7 to -68.8]
  12 Months: number analyzed (Participants) | 174 | 182
  12 Months | -69.3 [-73.7 to -65] | -73.8 [-78 to -69.6]

3. Secondary Outcome: Change From Baseline UDI Irritative Score
Description: The Urogenital Distress Inventory is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI Irritative subscale has a range from 0 to 100 with higher scores indicating greater distress. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 196
  3 Months | -49.7 [-53.3 to -46.2] | -50.1 [-53.6 to -46.6]
  6 Months: number analyzed (Participants) | 176 | 183
  6 Months | -49.5 [-53.2 to -45.7] | -53.5 [-56.9 to -50.1]
  12 Months: number analyzed (Participants) | 174 | 182
  12 Months | -50 [-53.6 to -46.4] | -53.5 [-57.1 to -49.9]

4. Secondary Outcome: Change From Baseline UDI Obstructive Score
Description: The Urogenital Distress Inventory is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI Obstructive subscale has a range from 0 to 100 with higher scores indicating greater distress. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 196
  3 Months | -18.5 [-20.9 to -16] | -20.2 [-23.4 to -16.9]
  6 Months: number analyzed (Participants) | 176 | 183
  6 Months | -18 [-20.6 to -15.4] | -21.1 [-24.2 to -18]
  12 Months: number analyzed (Participants) | 174 | 182
  12 Months | -18.5 [-21.1 to -15.9] | -20.3 [-23.7 to -17]

5. Other Pre Specified Outcome: Change From Baseline Number of Stress Incontinence Episodes
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in number of stress incontinence episodes at 2 weeks, 2, 6, or 12 months and the number of stress incontinence episodes at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of episodes
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -2.2 [-2.4 to -1.9] | -2.2 [-2.6 to -1.9]
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months | -2.3 [-2.6 to -2.1] | -2.4 [-2.7 to -2]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -2.3 [-2.6 to -2] | -2.3 [-2.6 to -2]
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months | -2.2 [-2.5 to -2] | -2.2 [-2.6 to -1.9]

6. Other Pre Specified Outcome: Change From Baseline Number of Urge Incontinence Episodes
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in number of urge incontinence episodes at 2 weeks, 2, 6, or 12 months and the number of urge incontinence episodes at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of episodes
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -1.8 [-2.2 to -1.5] | -1.7 [-2 to -1.4]
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months | -2 [-2.3 to -1.7] | -2 [-2.3 to -1.8]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -2 [-2.4 to -1.6] | -2 [-2.3 to -1.7]
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months | -1.9 [-2.3 to -1.5] | -2.2 [-2.5 to -1.8]

7. Other Pre Specified Outcome: Change From Baseline Number of Unknown Incontinence Episodes
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in number of unknown incontinence episodes at 2 weeks, 2, 6, or 12 months and the number of unknown incontinence episodes at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of episodes
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -0.2 [-0.3 to 0] | -0.4 [-0.5 to -0.2]
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months | -0.3 [-0.5 to -0.2] | -0.4 [-0.6 to -0.2]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -0.3 [-0.4 to -0.2] | -0.4 [-0.6 to -0.2]
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months | -0.3 [-0.4 to -0.1] | -0.4 [-0.6 to -0.2]

8. Other Pre Specified Outcome: Change From Baseline Total Number of Incontinence Episodes
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in total number of incontinence episodes at 2 weeks, 2, 6, or 12 months and the total number of incontinence episodes at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of episodes
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -4.2 [-4.7 to -3.7] | -4.3 [-4.8 to -3.8]
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months | -4.7 [-5.1 to -4.2] | -4.8 [-5.2 to -4.3]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -4.6 [-5.1 to -4.1] | -4.7 [-5.2 to -4.3]
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months | -4.4 [-4.9 to -3.9] | -4.8 [-5.3 to -4.3]

9. Other Pre Specified Outcome: Change From Baseline Number of Wet Pads Per Day
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in number of wet pads per day at 2 weeks, 2, 6, or 12 months and the number of wet pads per day at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of pads
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of pads
  0.5 Months: number analyzed (Participants) | 199 | 197
  0.5 Months | -2 [-2.3 to -1.7] | -2.2 [-2.6 to -1.8]
  2 Months: number analyzed (Participants) | 190 | 189
  2 Months | -2.4 [-2.7 to -2.1] | -2.7 [-3.1 to -2.2]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -2.2 [-2.6 to -1.8] | -2.7 [-3.1 to -2.2]
  12 Months: number analyzed (Participants) | 160 | 165
  12 Months | -2.2 [-2.6 to -1.9] | -2.7 [-3.1 to -2.2]

10. Other Pre Specified Outcome: Change From Baseline Number of Pads Per Day
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in total number of pads per day at 2 weeks, 2, 6, or 12 months and the total number of pads per day at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of pads
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of pads
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -1.6 [-1.9 to -1.3] | -1.9 [-2.3 to -1.5]
  2 Months: number analyzed (Participants) | 191 | 189
  2 Months | -2.2 [-2.6 to -1.9] | -2.7 [-3.1 to -2.2]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -2.2 [-2.6 to -1.8] | -2.8 [-3.3 to -2.3]
  12 Months: number analyzed (Participants) | 160 | 165
  12 Months | -2.3 [-2.7 to -2] | -2.7 [-3.2 to -2.3]

11. Other Pre Specified Outcome: Change From Baseline Number of Daytime Voids
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in number of daytime voids at 2 weeks, 2, 6, or 12 months and the number of daytime voids at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of voids
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of voids
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -0.6 [-1 to -0.3] | -0.8 [-1.2 to -0.4]
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months | -0.7 [-1 to -0.3] | -1.6 [-1.9 to -1.2]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -1.1 [-1.4 to -0.7] | -2.2 [-2.5 to -1.8]
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months | -1.2 [-1.6 to -0.8] | -2 [-2.4 to -1.7]

12. Other Pre Specified Outcome: Change From Baseline Number of Nighttime Voids
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in number of nighttime voids at 2 weeks, 2, 6, or 12 months and the number of nighttime voids at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of voids
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of voids
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -0.2 [-0.4 to -0.1] | -0.4 [-0.6 to -0.2]
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months | -0.4 [-0.6 to -0.3] | -0.7 [-0.8 to -0.5]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -0.5 [-0.7 to -0.4] | -0.8 [-0.9 to -0.6]
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months | -0.4 [-0.6 to -0.2] | -0.8 [-0.9 to -0.6]

13. Other Pre Specified Outcome: Change From Baseline Number of Urgency Voids Without Incontinence
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome variable is computed as the difference in number of urgency voids without incontinence at 2 weeks, 2, 6, or 12 months and the number of urgency voids without incontinence at baseline.
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of voids
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
number of voids
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months | -1.1 [-2.3 to 0.1] | -0.8 [-2.2 to 0.6]
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months | -1.6 [-3 to -0.3] | -4.3 [-5.8 to -2.8]
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months | -3.5 [-4.9 to -2.1] | -4.8 [-6.4 to -3.1]
  12 Months: number analyzed (Participants) | 159 | 165
  12 Months | -3.9 [-5.5 to -2.4] | -5.1 [-6.6 to -3.7]

14. Other Pre Specified Outcome: Number of Participants With <8 Voids After Baseline (Normalization of Voiding Frequency)
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, for participants with >8 voids at baseline, the outcome is calculated as Yes=no more than 8 voids noted at the time point, No=Otherwise
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
Participants
  0.5 Months: number analyzed (Participants) | 130 | 127
  0.5 Months: Yes | 48 | 59
  0.5 Months: No | 82 | 68
  2 Months: number analyzed (Participants) | 125 | 124
  2 Months: Yes | 49 | 81
  2 Months: No | 76 | 43
  6 Months: number analyzed (Participants) | 102 | 112
  6 Months: Yes | 46 | 79
  6 Months: No | 56 | 33
  12 Months: number analyzed (Participants) | 105 | 109
  12 Months: Yes | 48 | 80
  12 Months: No | 57 | 29

15. Other Pre Specified Outcome: Number of Participants With 50% Reduction in Voids Relative to Baseline (Improved Voiding Frequency)
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome is calculated as Yes=at least 50% reduction in the number of voids between 2 weeks, 2, 6, and 12 months and baseline, No=Otherwise
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
Participants
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months: Yes | 1 | 8
  0.5 Months: No | 198 | 190
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months: Yes | 2 | 13
  2 Months: No | 189 | 177
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months: Yes | 6 | 15
  6 Months: No | 152 | 155
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months: Yes | 8 | 15
  12 Months: No | 153 | 150

16. Other Pre Specified Outcome: Number of Participants With Greater Number of Voids Relative to Baseline or >8 Voids (Worsening Voiding Frequency)
Description: Based on data collected from participant-completed diaries at baseline, 2 weeks, and 2, 6, and 12 months, the outcome is calculated as Yes=greater than baseline number of voids at the time point or with greater than 8 voids at the time point, No=Otherwise
Time Frame: 2 weeks and 2, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
Participants
  0.5 Months: number analyzed (Participants) | 199 | 198
  0.5 Months: Yes | 124 | 104
  0.5 Months: No | 75 | 94
  2 Months: number analyzed (Participants) | 191 | 190
  2 Months: Yes | 111 | 68
  2 Months: No | 80 | 122
  6 Months: number analyzed (Participants) | 158 | 170
  6 Months: Yes | 81 | 43
  6 Months: No | 77 | 127
  12 Months: number analyzed (Participants) | 161 | 165
  12 Months: Yes | 79 | 43
  12 Months: No | 82 | 122

17. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSAPR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Not Partner Related subscale (NSA-PR) ranges from 0 to 100 with higher scores indicating worse function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 70 | 66
  3 Months | 7.1 [-0.8 to 15] | -8.8 [-16.6 to -1.1]
  6 Months: number analyzed (Participants) | 58 | 54
  6 Months | 5.5 [-2.9 to 13.8] | 2.5 [-7.6 to 12.6]
  12 Months: number analyzed (Participants) | 55 | 58
  12 Months | 3.3 [-6.9 to 13.6] | 2.3 [-5.8 to 10.4]

18. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSACS Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Not Sexually Active-Condition Specific subscale (NSA-CS) ranges from 0 to 100 with worse scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 65 | 60
  3 Months | -16.8 [-26.1 to -7.5] | -20.3 [-27.1 to -13.4]
  6 Months: number analyzed (Participants) | 53 | 50
  6 Months | -18.9 [-29.7 to -8] | -16.4 [-25.8 to -7.1]
  12 Months: number analyzed (Participants) | 51 | 53
  12 Months | -13.5 [-24.7 to -2.3] | -9.9 [-20.9 to 1.2]

19. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSAGQR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Not Sexually Active-Global Quality Rating subscale (NSA-GQR) ranges from 0 to 100 with higher scores indicating worse function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 66 | 61
  3 Months | -10 [-16.9 to -3.1] | -14.8 [-22.2 to -7.3]
  6 Months: number analyzed (Participants) | 54 | 49
  6 Months | -9.8 [-17.8 to -1.9] | -15.3 [-24.9 to -5.8]
  12 Months: number analyzed (Participants) | 51 | 53
  12 Months | -9.1 [-17.1 to -1] | -16.5 [-26 to -7]

20. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSACI Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Not Sexually Active-Condition Impact subscale (NSA-CI) ranges from 0 to 100 with higher scores indicating worse function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 67 | 61
  3 Months | -25.2 [-33.6 to -16.8] | -27.9 [-37.8 to -17.9]
  6 Months: number analyzed (Participants) | 54 | 49
  6 Months | -32.1 [-40.7 to -23.5] | -23.8 [-35.1 to -12.5]
  12 Months: number analyzed (Participants) | 52 | 53
  12 Months | -28.8 [-38.7 to -19] | -33 [-44.6 to -21.4]

21. Other Pre Specified Outcome: Change From Baseline PISQ-IR SAAO Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Sexually Active-Arousal, Orgasm subscale (SA-AO) ranges from 0 to 100 with higher scores indicating worse function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 101 | 103
  3 Months | 6.8 [3.7 to 9.9] | 10.8 [7.8 to 13.8]
  6 Months: number analyzed (Participants) | 88 | 98
  6 Months | 6.5 [2.9 to 10.1] | 12.1 [8.9 to 15.3]
  12 Months: number analyzed (Participants) | 92 | 102
  12 Months | 9.2 [6 to 12.4] | 9.6 [6.6 to 12.6]

22. Other Pre Specified Outcome: Change From Baseline PISQ-IR SAPR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Sexually Active-Partner Related subscale (SA-PR) ranges from 0 to 100 with higher scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 99 | 101
  3 Months | 5.2 [1.8 to 8.5] | 7 [3.1 to 11]
  6 Months: number analyzed (Participants) | 87 | 98
  6 Months | 4.9 [1.2 to 8.5] | 6.3 [2.1 to 10.6]
  12 Months: number analyzed (Participants) | 92 | 102
  12 Months | 2.3 [-1.7 to 6.3] | 4.6 [-0.3 to 9.5]

23. Other Pre Specified Outcome: Change From Baseline PISQ-IR SACS Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Sexually Active-Condition Specific subscale (SA-CS) ranges from 0 to 100 with higher scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 99 | 103
  3 Months | 21.1 [16.9 to 25.4] | 28.2 [23.3 to 33]
  6 Months: number analyzed (Participants) | 86 | 98
  6 Months | 20 [15.1 to 24.9] | 28.9 [23.7 to 34.1]
  12 Months: number analyzed (Participants) | 92 | 101
  12 Months | 24.2 [19.3 to 29.1] | 26.3 [21.6 to 31]

24. Other Pre Specified Outcome: Change From Baseline PISQ-IR SAGQR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Sexually Active-Global Quality Rating subscale (SA-GQR) ranges from 0 to 100 with higher scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 99 | 103
  3 Months | 13.5 [8.4 to 18.6] | 18.3 [13.5 to 23]
  6 Months: number analyzed (Participants) | 88 | 98
  6 Months | 12.1 [6.5 to 17.7] | 19 [14.1 to 24]
  12 Months: number analyzed (Participants) | 92 | 100
  12 Months | 19 [13.9 to 24.1] | 13.5 [7.9 to 19]

25. Other Pre Specified Outcome: Change From Baseline PISQ-IR SACI Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Sexually Active-Condition Impact subscale (SA-CI) ranges from 0 to 100 with higher scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 101 | 103
  3 Months | 28.4 [22.5 to 34.3] | 33.6 [27.6 to 39.5]
  6 Months: number analyzed (Participants) | 88 | 98
  6 Months | 28.9 [22.5 to 35.3] | 35.3 [28.9 to 41.7]
  12 Months: number analyzed (Participants) | 92 | 102
  12 Months | 31.7 [24.7 to 38.7] | 35.5 [29.4 to 41.7]

26. Other Pre Specified Outcome: Change From Baseline PISQ-IR SAD Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. Using the Rockwood scoring, the PISQ-IR Sexually Active-Desire subscale (SA-D) ranges from 0 to 100 with higher scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 101 | 103
  3 Months | 3.8 [0.8 to 6.9] | 7.1 [4.4 to 9.7]
  6 Months: number analyzed (Participants) | 88 | 98
  6 Months | 0.4 [-3.1 to 3.8] | 5.4 [2.7 to 8.1]
  12 Months: number analyzed (Participants) | 92 | 102
  12 Months | 2.7 [-0.7 to 6] | 2.5 [-0.8 to 5.7]

27. Other Pre Specified Outcome: Change From Baseline EQ-5D Index Score
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life. The index score ranges from 0 to 1 with higher scores indicating a better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 197 | 196
  3 Months | 0 [0 to 0.1] | 0 [0 to 0.1]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | 0 [0 to 0.1] | 0 [0 to 0.1]
  12 Months: number analyzed (Participants) | 174 | 181
  12 Months | 0 [0 to 0] | 0 [0 to 0.1]

28. Other Pre Specified Outcome: Change From Baseline EQ-5D Visual Analog Scale Score
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life. The visual analog scale (VAS) score ranges from 0 to 100 with higher scores indicating a better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 197 | 195
  3 Months | 0.3 [-2.5 to 3.1] | 4 [1 to 7]
  6 Months: number analyzed (Participants) | 176 | 180
  6 Months | 2.5 [-0.8 to 5.8] | 3.1 [-0.5 to 6.7]
  12 Months: number analyzed (Participants) | 173 | 180
  12 Months | 1.2 [-1.8 to 4.2] | 4.8 [1.6 to 7.9]

29. Other Pre Specified Outcome: Change From Baseline OABq-LF Symptom Severity Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Symptom Severity score ranges from 0 to 100 with higher score indicating worse quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 197 | 196
  3 Months | -45.3 [-48.7 to -41.8] | -46.9 [-50.2 to -43.7]
  6 Months: number analyzed (Participants) | 175 | 181
  6 Months | -45.4 [-49.2 to -41.6] | -47.2 [-50.8 to -43.6]
  12 Months: number analyzed (Participants) | 173 | 180
  12 Months | -45.7 [-49.6 to -41.8] | -48.5 [-52.2 to -44.8]

30. Other Pre Specified Outcome: Change From Baseline OABq-LF Coping Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Coping score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 196 | 197
  3 Months | 43.1 [39.1 to 47.1] | 48.2 [44.4 to 52]
  6 Months: number analyzed (Participants) | 175 | 182
  6 Months | 43.3 [38.9 to 47.6] | 48.4 [44.6 to 52.2]
  12 Months: number analyzed (Participants) | 173 | 181
  12 Months | 43.9 [39.6 to 48.2] | 47.9 [43.9 to 52]

31. Other Pre Specified Outcome: Change From Baseline OABq-LF Concern Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Concern score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 196 | 197
  3 Months | 47.6 [43.8 to 51.4] | 51.2 [47.2 to 55.1]
  6 Months: number analyzed (Participants) | 175 | 182
  6 Months | 47 [42.8 to 51.1] | 51.1 [47.3 to 54.9]
  12 Months: number analyzed (Participants) | 173 | 180
  12 Months | 46.9 [42.6 to 51.2] | 50.4 [46.4 to 54.5]

32. Other Pre Specified Outcome: Change From Baseline OABq-LF Sleep Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Sleep score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 196 | 197
  3 Months | 31.7 [27.8 to 35.6] | 31.6 [27.4 to 35.8]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | 31.3 [27.2 to 35.3] | 31.9 [27.5 to 36.3]
  12 Months: number analyzed (Participants) | 173 | 181
  12 Months | 31.8 [27.5 to 36.2] | 32.7 [28.1 to 37.3]

33. Other Pre Specified Outcome: Change From Baseline OABq-LF Social Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Social score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 197 | 197
  3 Months | 25.6 [21.8 to 29.4] | 26.5 [22.7 to 30.4]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | 23.5 [19.4 to 27.6] | 26.1 [22.2 to 30]
  12 Months: number analyzed (Participants) | 172 | 180
  12 Months | 24.1 [19.9 to 28.3] | 25.8 [21.8 to 29.9]

34. Other Pre Specified Outcome: Change From Baseline OABq-LF HRQL Total Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF HRQL score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 196 | 197
  3 Months | 38.6 [35.1 to 42] | 41.4 [37.9 to 44.8]
  6 Months: number analyzed (Participants) | 175 | 182
  6 Months | 38 [34.3 to 41.8] | 41.4 [38 to 44.8]
  12 Months: number analyzed (Participants) | 172 | 180
  12 Months | 38.6 [34.8 to 42.4] | 41.1 [37.4 to 44.8]

35. Other Pre Specified Outcome: OAB-SATq Satisfaction Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Satisfaction score ranges from 0 to 100 with higher scores indicating higher satisfaction.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 197 | 196
  3 Months | 19.3 [16 to 22.7] | 18.2 [15.2 to 21.3]
  6 Months: number analyzed (Participants) | 175 | 180
  6 Months | 19.8 [15.7 to 23.9] | 18.7 [15.3 to 22.2]
  12 Months: number analyzed (Participants) | 174 | 179
  12 Months | 18.1 [14.2 to 22.1] | 17.3 [14 to 20.6]

36. Other Pre Specified Outcome: OAB-SATq Side Effect Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Side Effect score ranges from 0 to 100 with higher scores indicating fewer side effects.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 195 | 196
  3 Months | 76 [70.6 to 81.3] | 84.3 [79.6 to 89]
  6 Months: number analyzed (Participants) | 174 | 181
  6 Months | 79.7 [74.3 to 85.1] | 87.2 [82.9 to 91.6]
  12 Months: number analyzed (Participants) | 174 | 179
  12 Months | 81 [75.7 to 86.4] | 86.3 [81.7 to 90.8]

37. Other Pre Specified Outcome: OAB-SATq Endorsement Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Endorsement score ranges from 0 to 100 with higher scores indicating greater endorsement.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 194 | 196
  3 Months | 10.6 [8.1 to 13] | 8.8 [6.5 to 11]
  6 Months: number analyzed (Participants) | 175 | 181
  6 Months | 11.2 [8 to 14.5] | 6.6 [4.5 to 8.7]
  12 Months: number analyzed (Participants) | 174 | 180
  12 Months | 10.7 [7.3 to 14] | 8.9 [6.5 to 11.4]

38. Other Pre Specified Outcome: OAB-SATq Convenience Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Convenience score ranges from 0 to 100 with higher scores indicating greater convenience.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 195 | 196
  3 Months | 18.8 [15.8 to 21.8] | 25.8 [22.8 to 28.9]
  6 Months: number analyzed (Participants) | 172 | 181
  6 Months | 19.1 [15.6 to 22.6] | 26.2 [22.8 to 29.6]
  12 Months: number analyzed (Participants) | 174 | 179
  12 Months | 19.7 [16 to 23.3] | 21.3 [18.1 to 24.6]

39. Other Pre Specified Outcome: OAB-SATq Preference Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The preference score is a binary [yes/no] indicator as to whether a subject indicated slight or definite preference for the treatment among women that have had previous treatment for overactive bladder. The outcome is the percentage of participants that prefer the current treatment to previous treatments.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
Participants
  3 Months: number analyzed (Participants) | 123 | 118
  3 Months: Yes | 111 | 109
  3 Months: No | 12 | 9
  6 Months: number analyzed (Participants) | 104 | 117
  6 Months: Yes | 101 | 112
  6 Months: No | 3 | 5
  12 Months: number analyzed (Participants) | 109 | 116
  12 Months: Yes | 98 | 107
  12 Months: No | 11 | 9

40. Other Pre Specified Outcome: Change From Baseline IIq-LF Physical Activity Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Physical Activity score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 196
  3 Months | -39.2 [-43.2 to -35.3] | -40.9 [-44.7 to -37.1]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | -39.1 [-43.5 to -34.8] | -42.1 [-46 to -38.1]
  12 Months: number analyzed (Participants) | 174 | 181
  12 Months | -42.3 [-46.3 to -38.3] | -42.5 [-46.5 to -38.4]

41. Other Pre Specified Outcome: Change From Baseline IIq-LF Travel Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Travel score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 196
  3 Months | -33.9 [-38.1 to -29.8] | -38.9 [-43.1 to -34.8]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | -33.4 [-38 to -28.8] | -40.9 [-45.3 to -36.5]
  12 Months: number analyzed (Participants) | 174 | 181
  12 Months | -35.4 [-39.9 to -30.9] | -40.8 [-45.1 to -36.4]

42. Other Pre Specified Outcome: Change From Baseline IIq-LF Social Relationship Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Social Relationship score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 196
  3 Months | -28.9 [-32.4 to -25.5] | -32.8 [-36.4 to -29.1]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | -28.6 [-32.4 to -24.9] | -33.7 [-37.4 to -30.1]
  12 Months: number analyzed (Participants) | 174 | 181
  12 Months | -30 [-33.8 to -26.1] | -34.1 [-37.9 to -30.2]

43. Other Pre Specified Outcome: Change From Baseline IIq-LF Emotional Health Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Emotional Health score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 196
  3 Months | -38.4 [-42.2 to -34.5] | -40.7 [-44.5 to -36.9]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | -38.6 [-42.6 to -34.5] | -41.5 [-45.2 to -37.8]
  12 Months: number analyzed (Participants) | 174 | 181
  12 Months | -38.3 [-42.4 to -34.3] | -42.8 [-46.7 to -39]

44. Other Pre Specified Outcome: Change From Baseline IIq-LF Total Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Total score ranges from 0 to 400 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 198 | 196
  3 Months | -140.4 [-154.2 to -126.7] | -153.3 [-167.3 to -139.3]
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months | -139.8 [-154.9 to -124.6] | -158.2 [-172.3 to -144.1]
  12 Months: number analyzed (Participants) | 174 | 181
  12 Months | -146 [-160.8 to -131.2] | -160.1 [-174.5 to -145.8]

45. Other Pre Specified Outcome: Change From Baseline ADI Hygiene Score
Description: The Adaptation Index is a standardized measure of health-related quality of life. The ADI Hygiene score ranges from 0 to 100 with higher score indicating worse severity in adaptive behaviors. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 193 | 196
  3 Months | -32.1 [-35.5 to -28.8] | -36.7 [-40 to -33.3]
  6 Months: number analyzed (Participants) | 172 | 180
  6 Months | -34.6 [-38.2 to -30.9] | -37.6 [-41 to -34.3]
  12 Months: number analyzed (Participants) | 170 | 177
  12 Months | -35.5 [-39.2 to -31.8] | -38.8 [-42.3 to -35.4]

46. Other Pre Specified Outcome: Change From Baseline ADI Avoidance Score
Description: The Adaptation Index is a standardized measure of health-related quality of life. The ADI Avoidance score ranges from 0 to 100 with higher score indicating worse severity in adaptive behaviors. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  3 Months: number analyzed (Participants) | 195 | 196
  3 Months | -31.3 [-34.7 to -27.8] | -33.8 [-37.1 to -30.6]
  6 Months: number analyzed (Participants) | 174 | 180
  6 Months | -32.5 [-36.1 to -28.8] | -34.5 [-38 to -30.9]
  12 Months: number analyzed (Participants) | 172 | 178
  12 Months | -33 [-36.8 to -29.2] | -35.7 [-39.2 to -32.2]

47. Other Pre Specified Outcome: Change From Baseline Brink Score
Description: The Brink scale considers three pelvic floor muscle contraction variables: vaginal pressure or muscle force, elevation or vertical displacement of the examiner fingers, and duration of contraction. The score ranges from 3 to 12 with higher scores indicating greater PFM function. The change from baseline outcome is calculated as the difference in score at 3 or 12 months and the score at baseline.
Time Frame: 2 weeks and 2 and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
units on a scale
  0.5 Months: number analyzed (Participants) | 214 | 198
  0.5 Months | 0.5 [0.2 to 0.8] | 0.2 [-0.1 to 0.6]
  2 Months: number analyzed (Participants) | 200 | 196
  2 Months | 0.5 [0.2 to 0.8] | 0.6 [0.3 to 0.9]
  12 Months: number analyzed (Participants) | 166 | 167
  12 Months | 0.6 [0.2 to 1] | 0.6 [0.3 to 1]

48. Other Pre Specified Outcome: Change From Average Peak Muscle Contraction Pressure (cm H2O)
Description: The average peak muscle contraction is measured during a physical exam. The outcome is calculated as the difference in measured value at 3 or 12 months and the score at baseline.
Time Frame: 2 weeks and 2 and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm H2O
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
cm H2O
  0.5 Months: number analyzed (Participants) | 201 | 180
  0.5 Months | 3.7 [1.8 to 5.6] | 0.7 [-1.3 to 2.7]
  2 Months: number analyzed (Participants) | 193 | 185
  2 Months | 5 [2.6 to 7.4] | 4.6 [1.9 to 7.3]
  12 Months: number analyzed (Participants) | 158 | 160
  12 Months | 4 [1.9 to 6.2] | 4.4 [1.5 to 7.2]

49. Other Pre Specified Outcome: PGI-I
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had improvement as indicated by a rating of 1 (very much better), 2 (much better).
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
Participants
  3 Months: number analyzed (Participants) | 197 | 197
  3 Months: Improved | 179 | 178
  3 Months: No Improvement/Worsened | 18 | 19
  6 Months: number analyzed (Participants) | 175 | 181
  6 Months: Improved | 156 | 168
  6 Months: No Improvement/Worsened | 19 | 13
  12 Months: number analyzed (Participants) | 174 | 181
  12 Months: Improved | 147 | 159
  12 Months: No Improvement/Worsened | 27 | 22

50. Other Pre Specified Outcome: PGI-S
Description: The Patient Global Impression of Severity (PGI-S) is a patient-reported measure of perceived severity of condition, as assessed on a scale of 1 (Normal) to 4 (Severe). Included here are participants who reported Normal or Mild severity as indicated by a rating of 1 or 2.
Time Frame: Baseline 3, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MUS Only | MUS+BPTx
Number analyzed (Participants) | 229 | 235
Participants
  0 Months: Normal/Mild | 41 | 48
  0 Months: Moderate/Severe | 188 | 187
  3 Months: number analyzed (Participants) | 197 | 198
  3 Months: Normal/Mild | 171 | 174
  3 Months: Moderate/Severe | 26 | 24
  6 Months: number analyzed (Participants) | 176 | 182
  6 Months: Normal/Mild | 155 | 166
  6 Months: Moderate/Severe | 21 | 16
  12 Months: number analyzed (Participants) | 174 | 180
  12 Months: Normal/Mild | 155 | 164
  12 Months: Moderate/Severe | 19 | 16

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | MUS Only | MUS+BPTx
All-Cause Mortality (participants affected / at risk) | 0/238 | 0/242
Serious Adverse Events (participants affected / at risk) | 28/238 | 21/242
Other Adverse Events (participants affected / at risk) | 163/238 | 172/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MUS Only (N=238) | MUS+BPTx (N=242)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bladder neck suspension (Surgical and medical procedures) | 2 (2) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
High frequency ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Tendon operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MUS Only (N=238) | MUS+BPTx (N=242)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Argininosuccinate lyase deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 2 (2) | 0 (0)
Blepharochalasis (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Pinguecula (Eye disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (13) | 11 (13)
Abdominal pain lower (Gastrointestinal disorders) | 5 (5) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (9) | 14 (16)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 7 (7)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 2 (2)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 1 (1)
Levator syndrome (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (8) | 4 (5)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 5 (5) | 4 (4)
Chills (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Hernia pain (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 2 (2) | 4 (4)
Oedema peripheral (General disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2)
Polyp (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic oedema (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 4 (4)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 4 (4)
Balanitis candida (Infections and infestations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 3 (3)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 4 (4) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 8 (9) | 1 (2)
Furuncle (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (3) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1)
Infected bunion (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 4 (4)
Nail bed infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 3 (3)
Otitis externa (Infections and infestations) | 2 (3) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 8 (9) | 8 (8)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 7 (7)
Urinary tract infection (Infections and infestations) | 60 (75) | 58 (74)
Vaginal infection (Infections and infestations) | 1 (1) | 5 (5)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 2 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 3 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to allergen (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anti-thyroid antibody (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 2 (2)
Blood thyroid stimulating hormone increas (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Cardiovascular function test abnormal (Investigations) | 0 (0) | 1 (1)
Erythrocytes sedimentation rate increased (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 2 (2) | 0 (0)
Helicobacter test positive (Investigations) | 0 (0) | 2 (2)
Prealbumin abnormal (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 18 (24)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 18 (20)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc annular tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (6)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11) | 8 (9)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Femoral nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 9 (10)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 4 (4) | 3 (4)
Morton's neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Resting tremor (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 6 (6)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 5 (5) | 0 (0)
Grief reaction (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 7 (7)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 3 (3) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 5 (5) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 1 (1) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 16 (16) | 17 (18)
Adnexa uteri mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Bartholin's cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 13 (13) | 11 (11)
Genital pain (Reproductive system and breast disorders) | 15 (15) | 4 (4)
Labia enlarged (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovulation pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 6 (7)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 6 (6) | 8 (8)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulva cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 5 (5)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (6)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Bartholin's cyst removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Foot operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 1 (1)
Tympanoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Vaginectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-02-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT01959347/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT01959347/SAP_001.pdf